CLINICAL TRIAL: NCT06698029
Title: Optimisation du Ciblage du VIM Pour la Radiochirurgie Dans le Tremblement sévère
Brief Title: Optimizing VIM Targeting for Radiosurgery in Severe Tremor
Acronym: OptiRS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCAPHM23_0448
Record Dates: First submitted 2024-06-24; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-06

CONDITIONS: Tremor; Laser Therapy
MeSH Terms: conditions — Tremor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the primary endpoint will be assessed at one year, in a blinded,manner
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIM radiosurgery with RebrAIn targeting technique (Experimental): VIM radiosurgery with RebrAIn targeting technique (model VIM-RS-LAT-1.0)
  Interventions: Other: VIM Targeting
- VIM radiosurgery standard targeting technique (No Intervention): VIM radiosurgery standard targeting technique

INTERVENTIONS:
Other: VIM Targeting — Targeting with the use of VIMRS-LAT-1.0
  Arms: VIM radiosurgery with RebrAIn targeting technique

SUMMARY:
Essential tremor is a common neurological disease, the most severe form of which combines postural and intention tremor, with significant physical, psychological and social repercussions. It is in these most severe forms that surgical lesioning of the ventro-intermediate nucleus of the thalamus (VIM) has been proposed. The VIM and its region of interest are almost impossible to identify directly on imaging (especially MRI), as it is part of the thalamus, which has the same intensity. To identify it, teams use average coordinates from stereotactic atlases (imprecise due to the high inter-individual variability of brain anatomy) or retrospective series of implanted patients. The hypothesis of the present trial is that the VIM-RS-LAT-1.0 algorithm developed by RebrAIn for radiosurgery will enable targeting that is at least as effective as conventional targeting. This is a single-center, controlled study, the primary endpoint of which will be assessed at one year, in a blinded, phase 3, comparative, non-inferiority, randomized study in two parallel groups of patients with severe tremor undergoing radiosurgery. In the control group, VIM will be targeted conventionally, and in the experimental group, VIM will be targeted by the RebrAIn algorithm (VIM-RS-LAT-1.0 model) of radiosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, disabling, drug-resistant essential tremor
* Patient selected as part of the multidisciplinary concertation meeting on abnormal movements
* Patient aged 18 to 85
* Brain MRI showing no anatomical abnormality contraindicating radiosurgical procedure
* MATTIS ≥ 130
* Subject affiliated to or benefiting from a social security scheme
* Free, informed and written consent signed by the participant and the investigator (no later than the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patients with a contraindication to brain MRI (pacemaker, intracerebral metal object, etc.)
* Pregnant or breast-feeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage improvement in tremor in the treated upper limb | between inclusion and one year post-operatively (after radiosurgery)
  Assessed on a composite tremor assessment criterion that strictly replicates the endpoint of the prospective study. The percentage will be considered as a continuous variable, between 0 and 100%, and will be assessed blindly by a single practitioner.

SECONDARY OUTCOMES:
The percentage of improvement in quality of life | Between inclusion and one year post-operatively (after radiosurgery)
  QUEST scale
Assessment of % change in postural balance | Between inclusion and one year post-operatively (after radiosurgery)
  SARA scale
Assessment of tolerability | At 12 months
  Surgical complications: permanent or non-permanent neurological complications assessed by clinical examination
Assessment of cognitive performance | At one year postradiosurgery
  Score of Mattis Dementia Rating Scale and the Verbal Fluency Test
Assess lesion location in relation to targeting | 12 months after radiosurgery
  MRI
Medico-economic evaluation of automatic targeting compared with conventional targeting | 12 months after radiosurgery
  QALY and EQ5D-5L scores

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided